

### STATISTICAL ANALYSIS PLAN

Protocol Number: TAV-ONYC-401

Title: An Open-label Study to Evaluate the Safety, Tolerability, and

Pharmacokinetics of KERYDIN<sup>®</sup> (tavaborole) topical solution, 5% in the Treatment of Onychomycosis of the Toenail in Pediatric

Subjects Ages 6 to 16 Years and 11 Months

Study Phase: 4

Expected Sample Size: Approximately 40 subjects

Sponsor: Anacor Pharmaceuticals, Inc.

1020 East Meadow Circle Palo Alto, CA 94303

Sponsor Representative: PPD , PhD

PPD

Statistician: PPD , PhD

QST Consultations, Ltd. 11275 Edgewater Drive Allendale, MI 49401

PPD

Protocol Version: Amendment 3, 28 March 2016

SAP Version / Date: Version 1 / September 13, 2016

Version 2 / June 2, 2017

Prepared by: PPD MS

**QST** Consultations, Ltd.

### APPROVAL STUDY TITLE: Protocol TAV-ONYC-401: An Open-label Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of KERYDIN® (tavaborole) topical solution, 5% in the Treatment of Onychomycosis of the Toenail in Pediatric Subjects Ages 6 to 16 Years and 11 Months I approve the Statistical Analysis Plan, Version 2, dated June 1, 2017. SIGNATURE: \_ DATE PPD PRPS., MBA AFFILIATION: QST Consultations, Ltd. PPD PPD SIGNATURE: DATE PPD , PhD AFFILIATION: Anacor Pharmaceuticals, Inc.

Revisions to the Statistical Analysis Plan described herein must be approved through a formal written amendment with the exception of minor editorial changes to tables, figures, or listing shells, and any necessary textual clarifications for programmers that do not affect the stated analysis variables, study endpoints, or statistical methods.

# **Change History:**

Table numbers were updated.

Table 14.4.2 Summary of Concomitant Medications was added.

No other changes were made to the statistical methods.

# 1. TABLE OF CONTENTS

| 1. | TA | BLE O | F CONTEN | NTS | 4 |
|---|---|---|---|---|---|
| 2. | LIS | ST OF A | BBREVIA | TIONS AND DEFINITIONS OF TERMS | 6 |
| 3. | INT | Γ <b>RODU</b> | CTION | | 7 |
| 4. | | | | S | |
| <b>5.</b> | | | | _ PLAN | |
| | 5.1 | | | sign | |
| | | 5.1.1 | | of Visits and Assessments | |
| | 5.2 | Selecti | ion of Study | Population | 10 |
| | | 5.2.1 | | Criteria | |
| | | 5.2.2 | | ı Criteria | |
| | 5.3 | Treatn | | | |
| | 5.4 | | | ty Variables | |
| | | 5.4.1 | • | Variables | |
| | | | 5.4.1.1 | | |
| | | | 5.4.1.2 | KOH Mount and Central Fungal Culture | 12 |
| | | 5.4.2 | Pharmaco | okinetic Assessments | 13 |
| | | 5.4.3 | Safety Va | riables | 13 |
| | | | 5.4.3.1 | Local Tolerability Reactions | 13 |
| | | | 5.4.3.2 | Vital Signs | |
| | | | 5.4.3.3 | Clinical Safety Laboratory Parameters and Pregnancy Tests | |
| | | | 5.4.3.4 | Adverse Events | 16 |
| | 5.5 | Statist | ical Method | s | 16 |
| | | 5.5.1 | Dispositio | on of Patients | 16 |
| | | 5.5.2 | | Analyzed | |
| | | 5.5.3 | | phic and Other Baseline Characteristics | |
| | | | 5.5.3.1 | Concomitant Medications | 17 |
| | | 5.5.4 | Measuren | nents of Treatment Compliance | 17 |
| | | 5.5.5 | Analysis | of Efficacy | 17 |
| | | 5.5.6 | Statistical | /Analytical Issues | 18 |
| | | | 5.5.6.1 | Adjustments for Covariates | 18 |
| | | | 5.5.6.2 | Handling of Dropouts or Missing Data | |
| | | | 5.5.6.3 | Interim Analyses and Data Monitoring | |
| | | | 5.5.6.4 | Multicenter Studies | |
| | | | 5.5.6.5 | Multiple Comparisons/Multiplicity | 18 |

| | | | 5.5.6.6 | Use of an "Efficacy Subset" of Patients | 18 |
|---|---|---|---|---|---|
| | | | 5.5.6.7 | Active-Control Studies Intended to Show Equivalence | 18 |
| | | | 5.5.6.8 | Examination of Subgroups | 18 |
| | | 5.5.7 | Pharmaco | okinetics | 18 |
| | | 5.5.8 | Safety A | nalyses | 19 |
| | | | 5.5.8.1 | Extent of Exposure | 19 |
| | | | 5.5.8.2 | Adverse Events | 19 |
| | | | 5.5.8.3 | Local Skin Reactions | 20 |
| | | | 5.5.8.4 | Safety Laboratory Values | 20 |
| | | | 5.5.8.5 | Vital Sign Measurements | 20 |
| | | 5.5.9 | Determin | nation of Sample Size | 20 |
| | 5.6 | Chang | es in the Pl | anned Analyses | 20 |
| 6. | INI | DEX OF | PLANNE | D END-OF-TEXT TABLES | 21 |
| 7. | INI | DEX OF | FPLANNE | D LISTINGS | 68 |

### 2. LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS

AE Adverse event

AUC $_{0-24}$  Area Under the plasma Concentration-time curve from Hour 0 to Hour 24 AUC $_{0-\infty}$  Area Under the plasma Concentration-time curve from Hour 0 extrapolated

to infinity

CN Clear Nail

C<sub>max</sub> maximum observed plasma concentration

CRF Case report form

DSO Distal subungal onychomycosis

MedDRA Medical Dictionary for Regulatory Affairs

 $\lambda_Z$  elimination rate constant LTR Local Tolerability Reactions

NSample sizePKPharamacokineticSAESerious adverse eventSDStandard deviation $t_{1/2}$ elimination half-life

TEAE Treatment-emergent adverse event

TGT Target great toenail

T<sub>max</sub> time to maximum observed plasma concentration

UPT Urine Pregnancy Test
WHO World Health Organization

### 3. INTRODUCTION

KERYDIN® (tavaborole) topical solution, 5%, the first oxaborole antifungal agent, was approved by the Food and Drug Administration for the topical treatment of onychomycosis of the toenails on 07 July 2014 (NDA 204427). This protocol is intended to satisfy the post-marketing study requirements (PMR-2154-1) and the Written Request of KERYDIN (tavaborole) topical solution, 5% in pediatric subjects with onychomycosis of the toenails.

### 4. STUDY OBJECTIVES

The primary objective of this study is to assess the safety and tolerability of KERYDIN (tavaborole) topical solution, 5% applied once daily for 48 weeks in pediatric subjects ages 6 to 16 years and 11 months with onychomycosis of the toenails.

The secondary objective is to perform PK assessments in a subgroup of at least 16 evaluable subjects ages 12 to 16 years and 11 months following topical administration under maximal use conditions.

### 5. INVESTIGATIONAL PLAN

### 5.1 Overall Study Design

This is an open-label study to evaluate the safety, tolerability, and pharmacokinetics of KERYDIN (tavaborole) topical solution, 5% in treating distal subungal onycomychosis (DSO) of the toenail in pediatric subjects ages 6 to 16 years and 11 months. An eligible subject will have a target great toenail (TGT) with at least 20% involvement with a positive potassium hydroxide (KOH) wet mount and positive fungal culture for *T. rubrum* or *T. mentagrophytes* from a sample obtained from an affected great toenail during the Screening period. KOH and fungal culture will be sent to a central mycology laboratory for eligibility determination. Both great toenails can be sampled at Screening.

The mycological confirmation of eligibility will be performed as follows:

- 1. Initial sample is KOH (+) and culture (+) for *T. rubrum* or *T. mentagrophytes*, with or without co-infection with *Candida* spp. or *E. floccosum*, subject is eligible for enrollment within the maximum period of 10 weeks (i.e., within 70 days) from the Screening visit.
- 2. Initial sample is KOH (-) or initial sample is KOH (+) and culture (-): The sample may be repeated and will be assessed as follows:
  - If a repeat sample is KOH (+) and culture (+) for *T. rubrum* or *T. mentagrophytes* with or without co-infection with *Candida* spp. or *E. floccosum*, for enrollment as long as the subject is enrolled within the maximum period of 10 weeks (i.e., within 70 days) from the Screening visit.

Eligible subjects will apply KERYDIN (tavaborole) topical solution, 5% once daily to all affected toenails (the TGT as well as all other toenails identified by the Investigator at the Baseline visit as having the clinical characteristics of onychomycosis) throughout the 48-week treatment period.

Subjects will be evaluated at Screening, Baseline (Day 1), and at Weeks 2, 4, 8, 16, 24, 32, 40, 48, and 52. Each evaluation will include a clinical assessment of the adverse events (AEs) and local tolerability evaluation.

Additional procedures are performed as follows:

- Mycology sampling at Screening, Week 24, and Week 52/early termination (ET)
- Clinical disease severity of the TGT at Screening, Week 24, and Week 52/ET
- Safety laboratory testing at Baseline, Week 24, and Week 52/ET
- Digital photography at Screening, Week 24, and Week 52/ET
- Urine pregnancy tests (UPTs) will be performed on all postmenarchal females at all scheduled visits starting at the Baseline visit.

Subjects will start diaries at Baseline (Day 1) and will complete the diary as instructed.

In this study, there will be a PK subgroup of at least 16 evaluable subjects ages 12 to 16 years and 11 months studied under maximal use conditions. Subjects in this maximal use subgroup will apply the study drug on all 10 toenails, including up to 2 mm of the surrounding skin, for 28 days (±7 days). On Day 15, a pre-dose PK sample will be collected to assess steady state trough level. On Day 29, the study drug application will be done at the study site, and PK samples will be collected prior to dosing, as well as 4, 6, 8, and 24 hours post-dose on Days 29-30. After PK sampling is complete, study drug will be applied only to the affected toenails.

### 5.1.1 Schedule of Visits and Assessments

| Study Visit No. | 1 | 2 | 3 | 4 | 4a | 5 | 6 | 7 | 8 | 9 | 10 | 11 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Visit 140. | (Screenin | (Baseli | | - | (P | | | • | | | 10 | (or |
| | <b>g</b> ) | ne) | | | K) | | | | | | | ÈT) |
| Study Day (±7 days V4-11, +7 | Up to -70 | ĺ | | | 30 | | | | | | | , |
| days V3) | days | 1 | 15 | 29 | | | | | | | | |
| Study Week | | | 2 | 4 | | 8 | 16 | 24 | 32 | 40 | 48 | 52 |
| Informed consent | X | | | | | | | | | | | |
| Obtain subject number | X | | | | | | | | | | | |
| Demographics | X | | | | | | | | | | | |
| Medical and medication history | X | X | | | | | | | | | | |
| Abbreviated physical | | X | | | | | | | | | | |
| examination | | | | | | | | | | | | |
| KOH mount and fungal culture <sup>c</sup> | X | | | | | | | X | | | | X |
| Review inclusion/exclusion | X | X | | | | | | | | | | |
| criteria | | | | | | | | | | | | |
| Identify target great toenail | X | X | | | | | | | | | | |
| (TGT) | | | | | | | | | | | | |
| Identify 'other toes' to be treated | | X | | | | | | | | | | |
| Clinical assessment (% TGT | X | | | | | | | X | | | | X |
| disease severity) | | | | | | | | | | | | |
| Concomitant medications | X | X | X | X | X | X | X | X | X | X | X | X |
| Adverse events (AEs) | X | X | X | X | X | X | X | X | X | X | X | X |
| Safety laboratory tests | | X | | | | | | X | | | | X |
| Urine pregnancy test (UPT) for | | X | X | X | | X | X | X | X | X | X | X |
| postmenarchal females | | | | | | | | | | | | |
| Vital signs (blood pressure, | X | X | X | X | | X | X | X | X | X | X | X |
| pulse rate, respiratory rate) <sup>a</sup> | | | | | | | | | | | | |
| LTR assessment | | X | X | X | | X | X | X | X | X | X | X |
| PK subgroup sampling <sup>b</sup> | | | X | X | x <sup>b</sup> | | | | | | | |
| Photography of the TGT <sup>c</sup> | X | | | | | | | X | | | | X |
| Weigh and dispense new study | | X | X | X | | X | X | X | X | X | | |
| drug kit | | | | | | | | | | | | |
| Study drug | | | X | X | | X | X | X | X | X | X | |
| collection/weighing/accountabili | | | | | | | | | | | | |
| ty | | | | | | | | | | | | |
| Supervise study drug self- | | X | X | X | | X | X | X | X | X | | |
| administration <sup>d</sup> | | | | | | | | | | | | |
| Diary review and training/re- | | X | X | X | | X | X | X | X | X | X | |
| training | | | | | | | | | | | | |
| Schedule next visit | X | X | X | X | 1 .: | X | X | X | X | X | X | |

ET, early termination; KOH, potassium hydroxide; PK, pharmacokinetic; LTR, local tolerability reaction

<sup>&</sup>lt;sup>a</sup> Vital signs conducted after subject is sitting or supine for at least 5 minutes.

b For subjects in the PK subgroup, at Visit 3 (Day 15) a pre-dose sample will be collected and Visit 4 (Day 29), PK samples will be collected prior to dosing, as well as 4, 6, and 8 hours post-dose. At Visit 4a (Day 30), the 24-hour post-dose sample is collected prior to dosing.

<sup>&</sup>lt;sup>c</sup> Perform photography procedures before mycology procedures.

d Application occurs at the site on visit days. For PK subgroup participants, the application for Visit 3 (Day 15) and Visit 4a (Day 30) is to occur after the subject has had their PK specimen drawn.

### 5.2 Selection of Study Population

### 5.2.1 Inclusion Criteria

Subjects must meet all of the following inclusion criteria to be eligible for this study:

- 1. Male or female subjects, ages  $\geq$  6 years and  $\leq$  16 years and 11 months at the time of enrollment
- 2. Have a parent or guardian able to understand, to agree to, and to sign the study ICF; subject has the ability to give assent based on their age, maturity, and psychological state at the time of parental/guardian consent
- 3. A clinical diagnosis of DSO affecting either great toenail with positive KOH and *T. rubrum* or *T. mentagrophytes* culture from the TGT confirmed by a central mycology laboratory during the Screening period
- 4. DSO involving at least 20% of the TGT
- 5. TGT capable of growing, as assessed by the Investigator or qualified designee
- 6. Subject and parent/guardian (if applicable) are willing and able to comply with study drug instructions, comply with study instructions, and commit to attending all visits
- 7. Postmenarchal females must agree to use a medically accepted method of contraception for the entire study period

### 5.2.2 Exclusion Criteria

Subjects who meet any of the following exclusion criteria will be excluded from entering the study:

- 1. One or more of the following conditions affecting the TGT:
  - Proximal subungual onychomycosis
  - Onychomycosis involving the lunula
  - Superficial white onychomycosis, dermatophytoma, exclusively lateral disease, or yellow/brown spikes
  - Screening culture results that demonstrate co-infection with *Scopulariopsis* spp., *Scytalidium* spp. or other nondermatophyte molds (exception: *Candida* spp. and *E. floccosum* are permitted)

- 2. Anatomic abnormalities of the toe(s) or toenail(s) to be treated including, but not limited to: genetic nail disorders, pigmentary disorders, onychogryphosis, trauma to the toenail(s) to be treated, or other abnormality that in the Investigator's opinion may interfere with clinical evaluation of the toenail(s) or would indicate that the subject is unlikely to respond to a topical treatment for DSO
- 3. Current or past history of chronic moccasin-type tinea pedis (involving the sides or dorsum of the foot)
- 4. Current or past history of psoriasis or lichen planus involving the skin, nails or mucous membranes
- 5. History of any significant chronic fungal disease other than onychomycosis (eg, chronic mucocutaneous candidiasis)
- 6. Known diagnosis of type I or type II diabetes
- 7. Concurrent use of or have used any of the following topical or systemic medications within the indicated timeframe prior to Screening:
  - Topical antifungals applied to the toenails: 2 weeks
  - Systemic corticosteroids (including intramuscular injections): 4 weeks
  - Systemic immunosuppressive agents: 4 weeks
  - Systemic antifungals for treatment of onychomycosis or with known activity against dermatophytes: 24 weeks
- 8. Any significant active or past medical condition which, in the Investigator's opinion, may expose the subject to unacceptable risk by study participation, confound the evaluation of treatment response or AEs, or interfere with the subject's ability to complete the study
- 9. History of any known immunodeficiency
- 10. Known to be allergic to the study drug or excipients in the study drug
- 11. History of drug or alcohol abuse (current or within the past 6 months)
- 12. Participated in any other trial of an investigational drug or device within 30 days prior to Screening or participation in a research study concurrent with this study

### 5.3 Treatments

KERYDIN (tavaborole) topical solution, 5% will be applied topically once daily for 48 weeks.

### 5.4 Efficacy and Safety Variables

### 5.4.1 Efficacy Variables

The efficacy assessments are intended to assess compliance with treatment for the purposes of the safety assessment.

### 5.4.1.1 Clinical Assessment of the Target Toenail Involvement

Clinical involvement of the TGT will be assessed at Screening and Weeks 24 and 52/ET using the following definitions of disease severity:

- Completely CN: no clinical evidence of onychomycosis as evidenced by normal toenail plate, no onycholysis, and no subungual hyperkeratosis
- **Almost CN**: no more than minimal evidence of onychomycosis as evidenced by toenail plate dystrophic or discolored ≤ 5% of the distal aspect, with minimally evident onycholysis and subungual hyperkeratosis
- **Mild onychomycosis**: onychomycosis as evidenced by toenail plate dystrophic or discolored > 5% to ≤ 20% of the distal aspect, with clearly evident onycholysis and subungual hyperkeratosis
- Moderate onychomycosis: onychomycosis as evidenced by toenail plate dystrophic or discolored > 20% to ≤ 50% of the distal aspect, with clearly evident onycholysis and subungual hyperkeratosis
- **Severe onychomycosis**: onychomycosis as evidenced by a toenail plate dystrophic or discolored > 50% of the distal aspect, with pronounced onycholysis and subungual hyperkeratosis

### **5.4.1.2 KOH Mount and Central Fungal Culture**

Mycology sampling is to occur after all photography procedures for that visit have been completed. At Screening, the Investigator may perform a KOH wet mount at the study site to confirm the clinical diagnosis of onychomycosis prior to obtaining a sample for the central mycology laboratory; however, care must be taken to obtain sufficient subungual debris for the analysis at the central laboratory. The local KOH wet mount is an optional procedure and only the central mycology laboratory reading will be used for analysis and eligibility determination. If both great toenails are potentially eligible by clinical criteria, then both great toenails can be sampled at Screening. A subject that fails mycology criteria may be resampled.

A sample of subungual debris will be obtained again at Week 24 and Week 52/ET.

### **5.4.2** Pharmacokinetic Assessments

Blood samples for the determination of plasma levels of tavaborole and PK parameters will be obtained under maximal use conditions (once daily application to all 10 toenails, including up to 2 mm of the surrounding skin) from the subgroup of subjects ages 12 to 16 years and 11 months to achieve at least 16 evaluable subjects. Subjects in the maximal use subgroup will apply the study drug on all 10 toenails, including up to 2 mm of the surrounding skin, for 28 days ±7 days. At Visit 3 (Day 15) a pre-dose PK sample will be collected to assess steady state trough level. At Visit 4 (Day 29), the study drug application will be done at the study site, and PK samples will be collected prior to dosing, as well as 4, 6, and 8 hours post-dose. At Visit 4a (Day 30) the sample will be collected 24 hours post-dose and prior to the application for that day.

Approximately 24 mL of blood (6 samples, 4 mL each) will be taken from each of the 16 subjects for the PK determination.

### 5.4.3 Safety Variables

# **5.4.3.1** Local Tolerability Reactions

Safety evaluations will include local tolerability reactions (LTRs) (burning/stinging, induration/edema, oozing and crusting, pruritus, erythema, and scaling), as reported by the subject and/or evaluated by the Investigator at Baseline and each study visit thereafter. LTRs will be documented on the case report form (CRF) specifically designed to capture LTR information (local tolerability signs CRF) and not on the AE CRF. LTRs that require treatment (eg, with a concomitant medication or drug interruption or drug discontinuation) are an exception to this guideline; these LTRs should be documented on both the local tolerability signs CRF and on the AE CRF.

| Grade | Guideline |
|---|---|
| Burning/Stinging | • |
| 0 - None | No stinging/burning |
| 1 - Mild | Slight warm, tingling sensation; not really bothersome |
| 2 - Moderate | Definite warm; tingling/stinging sensation that is somewhat bothersome |
| 3 - Severe | Hot, tingling/stinging sensation that has caused definite discomfort |
| Induration/Edema | |
| 0 - None | No elevation |
| 1 - Mild | Barely perceptible elevation |
| 2 - Moderate | Clearly perceptible elevation but not extensive |
| 3 - Severe | Marked and extensive elevation |
| Oozing and Crustin | g |
| 0 - None | Absent |
| 1 - Mild | Faint signs of oozing |
| 2 - Moderate | Definite oozing or crust but with 5 or fewer sites per area |
| 3 - Severe | Marked and extensive oozing and crusting |
| Pruritus | · |
| 0 - None | No pruritus |
| 1 - Mild | Occasional, slight itching/scratching |
| 2 - Moderate | Constant or intermittent itching/scratching which is not disturbing sleep |
| 3 - Severe | Severe bothersome itching/scratching which is disturbing sleep |
| Erythema | • |
| 0 - None | No redness present |
| 1 - Mild | Faintly detectable erythema; very light pink |
| 2 - Moderate | Dull red, clearly distinguishable |
| 3 - Severe | Deep/dark red |
| Scaling | • |
| 0 - None | No scaling |
| 1 - Mild | Barely perceptible shedding, noticeable only on light scratching or rubbing |
| 2 - Moderate | Obvious but not profuse scaling |
| 3 - Severe | Heavy scale production |

#### 5.4.3.2 **Vital Signs**

Vital signs will be measured at each study visit after the subject has been sitting or supine for at least 5 minutes. Vital sign measurements taken will be blood pressure, pulse rate, and respiratory rate.

#### Clinical Safety Laboratory Parameters and Pregnancy Tests 5.4.3.3

Clinical safety laboratory parameters will be assessed at Baseline, Week 24, and Week 52/ET, if applicable. Laboratory tests may be repeated more often if clinically indicated. Blood samples may be taken with the subject in a non-fasting state.

All out-of-normal range laboratory values must be evaluated by the Investigator or subinvestigator as to whether they are clinically significant (i.e., require medical intervention or have clinical signs and/or symptoms). Abnormal clinical laboratory parameters that are considered clinically significant by the Investigator will be recorded on the AE CRF except Baseline visit. Clinically significant laboratory abnormalities noted from the Baseline visit will be recorded as medical history. The AE should be reported as a clinical diagnosis when possible. Laboratory tests will be performed by the central laboratory and are presented in Table 5.

UPTs will be performed at each scheduled visit on postmenarchal females starting at Baseline. If a UPT result is positive, the subject must be discontinued.

The Sponsor will designate a central laboratory for safety laboratory tests. All samples for clinical laboratory tests must be managed through the central laboratory designated by the Sponsor. Sample management (collection, storage, shipping, etc.) will be done according to the central laboratory instructions.

### **Safety Laboratory Parameters**

| Hematology | Chemistry |
|---|---|
| Hemoglobin | Blood urea nitrogen |
| Hematocrit | Creatinine |
| Red blood cell count | Glucose (nonfasting) |
| Platelet count | Sodium, Potassium |
| White blood cell count | Aspartate aminotransferase, alanine aminotransferase |
| Neutrophils | Total bilirubin |
| Eosinophils | Alkaline phosphatase |
| Monocytes | Albumin |
| Basophils | Total protein |
| Lymphocytes | Urine pregnancy test (all scheduled visits starting at Baseline) |

### **5.4.3.4** Adverse Events

An AE is any untoward medical occurrence or unintended change from the subject's Baseline (pretreatment) condition, including intercurrent illness, that occurs during a clinical trial after treatment has started, whether or not it is considered related to study treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of an investigational product.

An AE is meant to include events that are either new or represent detectable exacerbations of preexisting conditions, and does not imply any judgment about causality.

AEs will be assessed at each visit. Any AE occurring on or after the date of the dose of study drug administration on Day 1 and up to and including the completion/termination date will be counted as treatment-emergent.

Adverse experiences may include but are not limited to subjective or objective symptoms spontaneously reported by the subject and/or observed by the Investigator or medical staff, including laboratory abnormalities of clinical significance. Preexisting conditions noted as part of the medical history at Screening must be reported on the appropriate medical history CRF page. Stable, ongoing conditions present at Screening should not be recorded as AEs if the severity at Screening remains unchanged during the study. However, preexisting conditions for which an increase in severity is observed after Screening must be recorded as AEs.

### 5.5 Statistical Methods

All statistical processing will be performed using SAS® unless otherwise stated.

Descriptive statistics will include sample size, mean, median, standard deviation, minimum, and maximum continuous variables. Categorical variables will be tabulated with frequency counts and percentages.

### **5.5.1** Disposition of Patients

A tabulation of subject disposition will be provided. The tabulation will include the numbers of subjects who enter the study, complete the study, and discontinue the study. The reasons for discontinuation will be included.

### 5.5.2 Data Sets Analyzed

The following populations will be used:

• Safety population: all subjects who receive at least one confirmed dose of study drug and have at least one post-baseline safety assessment.

• **PK population:** all subjects from the maximal use subgroup with available PK data at Day 15 and at least one collection on Day 29.

### 5.5.3 Demographic and Other Baseline Characteristics

Subject demographic (age, sex, race, and ethnicity) and Baseline characteristics will be summarized for the Safety and PK populations. Age will be represented as both a continuous and as a categorical variable.

#### 5.5.3.1 Concomitant Medications

Concomitant medications will be coded using the World Health Organization Drug Dictionary Enhanced. All medications will be presented in the data listings. A table of concomitant medications by percentage of subjects who used them will also be provided. No statistical tests will be performed.

### 5.5.4 Measurements of Treatment Compliance

No formal evaluations of compliance are planned.

### 5.5.5 Analysis of Efficacy

Efficacy assessments will be summarized at Baseline, Week 24 and Week 52.

The primary efficacy endpoint for this study is the complete cure rate of the TGT at Week 52. Complete cure is defined as 0% clinical involvement of the TGT and negative mycology (negative KOH wet mount and negative fungal culture) at Week 52.

The secondary efficacy endpoints include the following:

- Complete or almost complete cure of the TGT at Weeks 24 and 52
- Treatment success (Clinical Efficacy rate) of the TGT at Weeks 24 and 52 defined as completely Clear Nail (CN) or almost CN
- Negative mycology (Mycological Cure rate) of the TGT at Weeks 24 and 52 defined as negative KOH wet mount and negative fungal culture
- Negative fungal culture of the TGT at Weeks 24 and 52

The primary and secondary efficacy endpoints will be summarized for the safety population with descriptive statistics including sample size, frequency count, and percentage.

### 5.5.6 Statistical/Analytical Issues

### **5.5.6.1** Adjustments for Covariates

No planned analyses include covariates.

### 5.5.6.2 Handling of Dropouts or Missing Data

No imputations will be made for missing data.

### 5.5.6.3 Interim Analyses and Data Monitoring

No interim analyses are planned.

### 5.5.6.4 Multicenter Studies

The study will be conducted at multiple investigational centers with the intention of pooling the results for analysis.

### 5.5.6.5 Multiple Comparisons/Multiplicity

Not applicable.

### 5.5.6.6 Use of an "Efficacy Subset" of Patients

Not applicable.

### 5.5.6.7 Active-Control Studies Intended to Show Equivalence

Not applicable.

### **5.5.6.8** Examination of Subgroups

No subgroup summaries are planned.

### 5.5.7 Pharmacokinetics

Pharmacokinetics will be tabulated for each collection day using descriptive statistics. Mean plasma concentrations will be plotted through time using both linear and semi-logarithmic scales. Plasma concentrations will also be plotted through time for each subject, using both linear and semi-logarithmic scales. Concentrations below the limit of quantitation will be set to zero for descriptive statistics.

The following PK parameters will be calculated for Day 15 (steady state trough level only) and Day 29 [steady state (±specified window)]:

• C<sub>max</sub>: maximum observed plasma concentration

• T<sub>max</sub>: time to maximum observed plasma concentration

• AUC<sub>0-24</sub>: area under the plasma concentration-time curve from Hour 0 to Hour 24, calculated using the linear trapezoidal rule

• AUC<sub>0- $\infty$ </sub>: area under the plasma concentration-time curve extrapolated to infinity

•  $\lambda_7$ : elimination rate constant

•  $t_{1/2}$ : elimination half-life

PK parameters will be calculated using actual sampling times.

### 5.5.8 Safety Analyses

No imputation will be made for missing safety data.

### 5.5.8.1 Extent of Exposure

The extent of exposure to study drug will be summarized by the total number of days of dosing, total number of applications, and total amount of study drug applied.

#### 5.5.8.2 Adverse Events

All AEs occurring during the study will be recorded and classified on the basis of *Medical Dictionary for Regulatory Activities* terminology. TEAEs are those with an onset on or after the time of the first study drug administration. For the safety population, all reported TEAEs will be summarized by system organ class (SOC), preferred term, severity, relationship to study drug, and seriousness. When summarizing TEAEs by causality and severity, each subject will be counted only once within an SOC or a preferred term using the event with the closest relationship to study drug and the greatest severity within each classification.

SAEs will be summarized by severity and relationship to study drug, and individual SAEs will be listed by subject. A list of subjects who prematurely discontinued from the study due to an AE will also be provided.

All information pertaining to AEs noted during the study will be listed by subject, detailing the verbatim term reported by the Investigator, preferred term, SOC, onset date, resolution date, maximum severity, seriousness, action taken regarding study drug, corrective treatment, outcome, and drug relationship. The event onset will also be shown relative (in number of days) to date of first administration of study drug.

### 5.5.8.3 Local Skin Reactions

LTRs (burning/stinging, induration/edema, oozing and crusting, pruritus, erythema, and scaling) will be evaluated by frequency tables for Baseline and Weeks 2, 4, 8, 16, 24, 32, 40, 48, and 52. Additionally, LTRs as well as change from baseline in LTRs will be summarized by descriptive statistics (mean, standard deviation, median, and minimum and maximum).

### 5.5.8.4 Safety Laboratory Values

Laboratory values as well as changes from Baseline in laboratory values will be summarized with descriptive statistics at Baseline, Week 24 and Week 52. In addition, shift tables will be created according to normal ranges. The last laboratory evaluation before the first dose of study drug will be used as Baseline for all laboratory analyses.

# 5.5.8.5 Vital Sign Measurements

Vital signs will be summarized with descriptive statistics at Baseline and Weeks 2, 4, 8, 16, 24, 32, 40, 48, and 52. Change from Baseline in vital signs will be summarized at Weeks 2, 4, 8, 16, 24, 32, 40, 48, and 52

### **5.5.9 Determination of Sample Size**

The study will enroll subjects ages 6 to 16 years and 11 months with at least 40 subjects ages 12 to 16 years and 11 months. All subjects will be assigned to receive active treatment with KERYDIN (tavaborole) topical solution, 5%. A PK subgroup of at least 16 evaluable subjects ages 12 to 16 years and 11 months will be studied under maximal use conditions.

The sample size is considered adequate to achieve the study objectives. No formal power calculations were performed.

### 5.6 Changes in the Planned Analyses

There are no changes to planned analyses. The PK population definition was clarified to include available PK data.

# 6. INDEX OF PLANNED END-OF-TEXT TABLES

| Table 14.1.1.1: Summary of Subject Completion/Discontinuation | 23 |
|---|---|
| Table 14.1.1.1: Summary of Subject Enrollment and Evaluability | 24 |
| Table 14.1.2.1: Summary of Subject Demographic Characteristics (Safety Population) | 25 |
| Table 14.1.2.2: Summary of Subject Demographic Characteristics (PK Population) | 26 |
| Table 14.1.2.3: Summary of Subject Baseline Characteristics (Safety Population) | 27 |
| Table 14.1.2.4: Summary of Subject Baseline Characteristics (PK Population) | 28 |
| Table 14.2.1: Summary of Clinical and Mycological Characteristics by Visit (Safety Population | on)29 |
| Table 14.2.2: Summary of the Primary Efficacy Endpoint: Complete Cure at Week 52 (Safety Population) | 30 |
| Table 14.2.3: Summary of Secondary Efficacy Endpoints (Safety Population) | 31 |
| Table 14.3.1.1.1: Summary of Local Tolerability Reactions by Visit (Safety Population) | 33 |
| Table 14.3.1.1.2: Means Summary of Local Tolerabilty Reactions by Visit (Safety Population) | )36 |
| Table 14.3.1.2.1: Summary of Treatment-Emergent Adverse Event Characteristics (Safety Population) | 42 |
| Table 14.3.1.2.2: Summary of Treatment-Emergent Adverse Events Leading to Permanent Withdrawal of Study Drug and/or Early Discontinuation From the Study (Safety Population) | 44 |
| Table 14.3.1.2.3: Summary of Treatment-Emergent Adverse Events by MedDRA System Org Class and Preferred Term (Safety Population) | |
| Table 14.3.1.2.4: Summary of Treatment-Emergent Adverse Events by Severity (Safety Population) | 46 |
| Table 14.3.1.2.4: Summary of Treatment-Emergent Adverse Events by Relationship (Safety Population) | 47 |
| Table 14.3.2.2.1: Summary of Treatment-Emergent Serious Adverse Event Characteristics (Safety Population) | 48 |
| Table 14.3.2.2.2: Summary of Treatment-Emergent Serious Adverse Events by MedDRA System Organ Class and Preferred Term (Safety Population) | 50 |
| Table 14.3.2.2.3: Summary of Treatment-Emergent Serious Adverse Events by Severity (Safety Population) | 51 |
| Table 14.3.2.2.4: Summary of Treatment-Emergent Serious Adverse Events by Relationship (Safety Population) | 52 |
| Table 14.3.4.1.1: Summary of Hematology Results (Safety Population) | 53 |
| Table 14.3.4.1.2: Summary of Chemistry Results (Safety Population) | 54 |
| Table 14.3.5.1: Summary of Vital Signs by Visit (Safety Population) | 55 |

| Table 14.4.1: Extent of Exposure (Safety Population) | 59 |
|---|---|
| Table 14.4.2: Summary of Concomitant Medications (Safety Population) | 60 |
| Table 14.4.4.1: Summary of Tavaborole Plasma Concentrations (PK Population) | 61 |
| Figure 14.4.4.1.1: Linear Plot of Mean Plasma Concentrations of Tavaborole by Time (PK Population) | 62 |
| Figure 14.4.4.1.2: Semi-logarithmic Plot of Mean Plasma Concentrations of Tavaborole by Time (PK Population) | 63 |
| Figure 14.4.4.1.3: By-Subject Linear Plots of Plasma Concentrations of Tavaborole by Time (P Population) | |
| Figure 14.4.4.1.4: By-Subject Semi-logarithmic Plots of Plasma Concentrations of Tavaborole by Time (PK Population) | |
| Table 14.4.5.1: Summary of Pharmacokinetic Parameters of Tavaborole at Day 29 (PK Population) | 66 |

Table 14.1.1.1: Summary of Subject Completion/Discontinuation

| | KERYDIN® |
|----------------------------|-----------------|
| | (N=xx) |
| Completed Study | |
| Yes | $XX (XX,X^0/6)$ |
| No | xx ( xx.x%) |
| Reason for Discontinuation | |
| Adverse Event | $XX (XX,X^{0})$ |
| Lost to Follow-Up | $xx(x^0/x)$ |
| Pregnancy | $xx(x^0/x)$ |
| Protocol Deviation | $XX (XX,X^0)$ |
| Withdrawal by Subject | $XX (XX,X^0)$ |
| Other | $XX (XX,X^0)$ |

Listing 16.2.1.1 SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table 14.1.1.1: Summary of Subject Enrollment and Evaluability

| | KERYDIN® |
|---------------------------------------------------------|----------|
| Number of Subjects Included in the Safety Population | XX |
| Number of Subjects Excluded from the Safety Population | XX |
| Reason for Exclusion from the Safety Population | |
| No Confirmed Dose of Study Drug | XX |
| No Post-Baseline Safety Assessment | XX |
| Number of Subjects Included in the Maximal Use Subgroup | XX |
| Number of Subjects Included in the PK Population | XX |
| Number of Subjects Excluded from the PK Population | XX |
| Reason for Exclusion from the PK Population | |
| Not Included in Maximal Use Subgroup | XX |
| No Available PK Data | XX |

Listing 16.2.3

Table 14.1.2.1: Summary of Subject Demographic Characteristics (Safety Population)

| | KERYDIN® |
|-------------------------------------------|-------------|
| | (N=xx) |
| Age (years) | |
| N | XX |
| Mean | XX.X |
| SD | XX.XX |
| Median | XX.X |
| Min. to Max. | xx to xx |
| 6 to less than 12 years | xx ( xx.x%) |
| 12 years to 16 years, 11 months | xx ( xx.x%) |
| Sex | |
| N | XX |
| Male | xx ( xx.x%) |
| Female | xx ( xx.x%) |
| Ethnicity | |
| N | XX |
| Hispanic or Latino | xx ( xx.x%) |
| Not Hispanic or Latino | xx ( xx.x%) |
| Race | |
| N | XX |
| American Indian or Alaska Native | xx ( xx.x%) |
| Asian | xx (xx.x%) |
| Black or African American | xx ( xx.x%) |
| Native Hawaiian or Other Pacific Islander | xx ( xx.x%) |
| White | xx (xx.x%) |

Listing 16.2.4.1

Table 14.1.2.2: Summary of Subject Demographic Characteristics (PK Population)

| | KERYDIN® |
|-------------------------------------------|-------------|
| | (N=xx) |
| Age (years) | (1\ AA) |
| N | XX |
| Mean | XX.X |
| SD | XX.XX |
| Median | XX.X |
| Min. to Max. | xx to xx |
| 6 to less than 12 years | xx ( xx.x%) |
| 12 years to 16 years, 11 months | $xx(x^{0})$ |
| Sex | |
| N | XX |
| Male | xx ( xx.x%) |
| Female | xx ( xx.x%) |
| Ethnicity | |
| N | XX |
| Hispanic or Latino | XX ( XX.X%) |
| Not Hispanic or Latino | xx ( xx.x%) |
| Race | |
| N | XX |
| American Indian or Alaska Native | xx ( xx.x%) |
| Asian | $xx(x^{2})$ |
| Black or African American | $xx(x^{2})$ |
| Native Hawaiian or Other Pacific Islander | xx ( xx.x%) |
| White | xx ( xx.x%) |

Listing 16.2.4.1

Table 14.1.2.3: Summary of Subject Baseline Characteristics (Safety Population)

| | KERYDIN® | |
|---|---|---|
| | (N=xx) | |
| Clinical Assessment of Disease Severity of Target Great Toenail | | _ |
| N | XX | |
| Completely Clear Nail | xx (xx.x%) | |
| Almost Clear Nail | xx (xx.x%) | |
| Mild Onychomycosis | xx (xx.x%) | |
| Moderate Onychomycosis | xx (xx.x%) | |
| Severe Onychomycosis | xx ( xx.x%) | |
| % Involvement of Target Great Toenail | | |
| N | XX | |
| Mean | XX.X | |
| SD | XX.XX | |
| Median | XX.X | |
| Min. to Max. | xx to xx | |
| Number of Other Affected Toenails | | |
| N | XX | |
| Mean | XX.X | |
| SD | XX.XX | |
| Median | XX.X | |
| Min. to Max. | xx to xx | |

Listings 16.2.6.1, 16.2.6.2

Table 14.1.2.4: Summary of Subject Baseline Characteristics (PK Population)

| | KERYDIN® | |
|---|---|---|
| | (N=xx) | |
| Clinical Assessment of Disease Severity of Target Great Toenail | , | _ |
| N | XX | |
| Completely Clear Nail | xx ( xx.x%) | |
| Almost Clear Nail | xx (xx.x%) | |
| Mild Onychomycosis | xx ( xx.x%) | |
| Moderate Onychomycosis | xx ( xx.x%) | |
| Severe Onychomycosis | xx ( xx.x%) | |
| % Involvement of Target Great Toenail | | |
| N | XX | |
| Mean | XX.X | |
| SD | XX.XX | |
| Median | XX.X | |
| Min. to Max. | xx to xx | |
| Number of Other Affected Toenails | | |
| N | XX | |
| Mean | XX.X | |
| SD | XX.XX | |
| Median | XX.X | |
| Min. to Max. | xx to xx | |

Listings 16.2.6.1, 16.2.6.2

Table 14.2.1: Summary of Clinical and Mycological Characteristics by Visit (Safety Population)

| KERYDIN® (N=xx) | Baseline | Week 24 | Week 52 |
|---|---|---|---|
| Clinical Assessment of Disease Severity of Target Grea | at | | |
| Toenail | | | |
| N | XX | XX | XX |
| Completely Clear Nail | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Almost Clear Nail | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Mild Onychomycosis | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Moderate Onychomycosis | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Severe Onychomycosis | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Fungal Culture Result ( <i>T. rubrum and T. mentagrophyt</i> | es) | | |
| N | XX | XX | XX |
| Positive | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Negative | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| KOH Result | | | |
| N | XX | XX | XX |
| Positive | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Negative | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

Note: No imputation of missing data.

Listing 16.2.6.1

Table 14.2.2: Summary of the Primary Efficacy Endpoint: Complete Cure at Week 52 (Safety Population)

| | KERYDIN®<br>(N=xx) |
|---------------------------------------|--------------------|
| Complete Cure <sup>a</sup> at Week 52 | , , |
| N | XX |
| Yes | xx ( xx.x%) |
| No | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Complete Cure defined as Completely Clear Nail, Negative Fungal Culture and Negative KOH.

Note: No imputation of missing data.

Listing 16.2.6.1

Table 14.2.3: Summary of Secondary Efficacy Endpoints (Safety Population) 

| | KERYDIN® |
|----------------------------------------------------------|-----------------|
| | (N=xx) |
| | (IV-XX) |
| Complete or Almost Complete Cure <sup>a</sup> at Week 24 | |
| N | XX |
| Yes | $XX (XX.X^{0})$ |
| No | xx (xx.x%) |
| Complete or Almost Complete Cure <sup>a</sup> at Week 52 | |
| N | XX |
| Yes | xx ( xx.x%) |
| No | xx ( xx.x%) |
| Treatment Success <sup>b</sup> at Week 24 | |
| N | XX |
| Yes | XX (XX.X%) |
| No | xx ( xx.x%) |
| Treatment Success <sup>b</sup> at Week 52 | |
| N | XX |
| Yes | xx ( xx.x%) |
| No | |
| INU | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Complete or Almost Complete Cure defined as Completely Clear or Almost Clear Nail, Negative Fungal Culture and Negative KOH.

<sup>b</sup> Treatment Success defined as Completely Clear or Almost Clear Nail.

<sup>c</sup> Negative Mycology defined as Negative Fungal Culture and Negative KOH.

Note: No imputation of missing data.

Listing 16.2.6.1

Table 14.2.3: Summary of Secondary Efficacy Endpoints (Safety Population) 

| | KERYDIN® |
|-------------------------------------------------------------|-------------|
| | (N=xx) |
| Negative Mycology <sup>c</sup> at Week 24 | |
| N | XX |
| Yes | xx (xx.x%) |
| No | xx ( xx.x%) |
| Negative Mycology <sup>c</sup> at Week 52 | |
| N | XX |
| Yes | xx ( xx.x%) |
| No | xx ( xx.x%) |
| Fungal Culture at Week 24 (T. rubrum and T. mentagrophytes) | |
| N | XX |
| Negative | xx (xx.x%) |
| Positive | XX ( XX.X%) |
| Fungal Culture at Week 52 (T. rubrum and T. mentagrophytes) | |
| N | XX |
| Negative | xx (xx.x%) |
| Positive | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Complete or Almost Complete Cure defined as Completely Clear or Almost Clear Nail, Negative Fungal Culture and Negative KOH.

<sup>b</sup> Treatment Success defined as Completely Clear or Almost Clear Nail.

<sup>c</sup> Negative Mycology defined as Negative Fungal Culture and Negative KOH.

Note: No imputation of missing data.

Listing 16.2.6.1

Table 14.3.1.1.1: Summary of Local Tolerability Reactions by Visit (Safety Population)


| VEDVDING (N) | | | | | |
|---|---|---|---|---|---|
| KERYDIN® (N=xx) Burning/Stinging | Baseline | Week 2 | Week 4 | Week 8 | Week 16 |
| N | XX | XX | XX | XX | XX |
| 0 – None | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 – Mild | XX (XX,X%) | XX (XX.X%)<br>XX (XX.X%) | xx ( xx.x%) | XX (XX.X%) | xx ( xx.x%) |
| 2 – Moderate | $\mathbf{x}\mathbf{x} (\mathbf{x}\mathbf{x}.\mathbf{x}\%)$ | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 – Severe | | ` / | 1 2.0 | | ` / |
| 3 – Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Week 24 | Week 32 | Week 40 | Week 48 | Week 52 |
| N | XX | XX | XX | XX | XX |
| 0 - None | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| 1 – Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 – Moderate | xx ( xx.x%) | xx (xx.x%) | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 – Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Induration/Edema | Baseline | Week 2 | Week 4 | Week 8 | Week 16 |
| N | XX | XX | XX | XX | XX |
| 0 – None | xx ( xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 1 – Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 – Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 – Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Week 24 | Week 32 | Week 40 | Week 48 | Week 52 |
| N | XX | XX | XX | XX | XX |
| 0 – None | xx ( xx,x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 – Mild | $\mathbf{x}\mathbf{x} \left( \mathbf{x}\mathbf{x}.\mathbf{x}\% \right)$ | xx (xx.x%) | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) |
| 2 – Moderate | XX (XX.X%) | XX (XX.X%) | xx ( xx.x%) | XX (XX.X%) | xx ( xx.x%) |
| 3 – Severe | 2 2 2 | 2 0/3 | 2 2/ | 2 2 ( | 2 0/ |
| 3 – 367616 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

Note: No imputation of missing data.

Listing 16.2.7.1

Table 14.3.1.1.1: Summary of Local Tolerability Reactions by Visit (Safety Population)


| VEDVNING (N-vv) | | | | | |
|---|---|---|---|---|---|
| KERYDIN® (N=xx) Oozing and Crusting | Baseline | Week 2 | Week 4 | Week 8 | Week 16 |
| N | XX | XX | XX | XX | XX |
| 0 – None | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 1 – Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| 2 – Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 – Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Week 24 | Week 32 | Week 40 | Week 48 | Week 52 |
| N | XX | XX | XX | XX | XX |
| 0 - None | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| 1 – Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 – Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 – Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Pruritus | Baseline | Week 2 | Week 4 | Week 8 | Week 16 |
| N | XX | XX | XX | XX | XX |
| 0 – None | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 – Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 – Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 – Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Week 24 | Week 32 | Week 40 | Week 48 | Week 52 |
| N | XX | XX | XX | XX | XX |
| 0 - None | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 – Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 – Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 – Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

Note: No imputation of missing data.

Listing 16.2.7.1

Table 14.3.1.1.1: Summary of Local Tolerability Reactions by Visit (Safety Population)


| VEDVDIN® (N-vv) | | | | | |
|---|---|---|---|---|---|
| KERYDIN® (N=xx) Erythema | Baseline | Week 2 | Week 4 | Week 8 | Week 16 |
| N | XX | XX | XX | XX | XX |
| 0 – None | xx (xx.x%) | xx ( xx.x%) | xx (xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| 1 – Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 – Moderate | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 – Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Week 24 | Week 32 | Week 40 | Week 48 | Week 52 |
| N | XX | XX | XX | XX | XX |
| 0 - None | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 1 – Mild | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 – Moderate | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 – Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Scaling | Baseline | Week 2 | Week 4 | Week 8 | Week 16 |
| N | XX | XX | XX | XX | XX |
| 0 - None | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 – Mild | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| 2 – Moderate | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| 3 – Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Week 24 | Week 32 | Week 40 | Week 48 | Week 52 |
| N | XX | XX | XX | XX | XX |
| 0 - None | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 1 – Mild | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 – Moderate | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 3 – Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

Note: No imputation of missing data.

Listing 16.2.7.1

Table 14.3.1.1.2: Means Summary of Local Tolerabilty Reactions by Visit (Safety Population)


| KERYDIN® (N=xx) | | | | | | |
|---|---|---|---|---|---|---|
| Burning/Stinging | Baseline | Week 2 | Week 4 | Week 8 | Week 16 | Week 24 |
| N | XX | XX | XX | XX | XX | XX |
| Mean | X.X | X.X | X.X | X.X | X.X | X.X |
| SD | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min. to Max. | x to x | x to x | x to x | x to x | x to x | x to x |
| Change from Baseline | | | | | | |
| N | | XX | XX | XX | XX | XX |
| Mean | | X.X | X.X | X.X | X.X | X.X |
| SD | | X.XX | X.XX | X.XX | X.XX | X.XX |
| Median | | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min. to Max. | | x to x | x to x | x to x | x to x | x to x |
| Burning/Stinging | | Week 32 | Week 40 | Week 48 | Week 52 | |
| N | | XX | XX | XX | XX | |
| Mean | | X.X | X.X | X.X | X.X | |
| SD | | X.XX | X.XX | X.XX | X.XX | |
| Median | | XX.X | XX.X | XX.X | XX.X | |
| Min. to Max. | | x to x | x to x | x to x | x to x | |
| Change from Baseline | | | | | | |
| N | | XX | XX | XX | XX | |
| Mean | | X.X | X.X | X.X | X.X | |
| SD | | X.XX | X.XX | X.XX | X.XX | |
| Median | | XX.X | XX.X | XX.X | XX.X | |
| Min. to Max. | | x to x | x to x | x to x | x to x | |

Note: No imputation of missing data.

Listing 16.2.7.1

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)
Table 14.3.1.1.2: Means Summary of Local Tolerabilty Reactions by Visit (Safety Population)


| KERYDIN® (N=xx) | | | | | | |
|---|---|---|---|---|---|---|
| nduration/Edema | Baseline | Week 2 | Week 4 | Week 8 | Week 16 | Week 2 |
| N | XX | XX | XX | XX | XX | XX |
| Mean | X.X | X.X | X.X | X.X | X.X | X.X |
| SD | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min. to Max. | x to x | x to x | x to x | x to x | x to x | x to x |
| Change from Baseline | | | | | | |
| N | | XX | XX | XX | XX | XX |
| Mean | | X.X | X.X | X.X | X.X | X.X |
| SD | | X.XX | X.XX | X.XX | X.XX | X.XX |
| Median | | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min. to Max. | | x to x | x to x | x to x | x to x | x to x |
| Induration/Edema | | Week 32 | Week 40 | Week 48 | Week 52 | |
| N | | XX | XX | XX | XX | |
| Mean | | X.X | X.X | X.X | X.X | |
| SD | | X.XX | X.XX | X.XX | X.XX | |
| Median | | XX.X | XX.X | XX.X | XX.X | |
| Min. to Max. | | x to x | x to x | x to x | x to x | |
| Change from Baseline | | | | | | |
| N | | XX | XX | XX | XX | |
| Mean | | X.X | X.X | X.X | X.X | |
| SD | | X.XX | X.XX | X.XX | X.XX | |
| Median | | XX.X | XX.X | XX.X | XX.X | |
| Min. to Max. | | x to x | x to x | x to x | x to x | |

Note: No imputation of missing data.

Listing 16.2.7.1

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table 14.3.1.1.2: Means Summary of Local Tolerabilty Reactions by Visit (Safety Population)


| KERYDIN® (N=xx) | | | | | | |
|---|---|---|---|---|---|---|
| Oozing and Crusting | Baseline | Week 2 | Week 4 | Week 8 | Week 16 | Week 24 |
| N | XX | XX | XX | XX | XX | XX |
| Mean | X.X | X.X | X.X | X.X | X.X | X.X |
| SD | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min. to Max. | x to x | x to x | x to x | x to x | x to x | x to x |
| Change from Baseline | | | | | | |
| N | | XX | XX | XX | XX | XX |
| Mean | | X.X | X.X | X.X | X.X | X.X |
| SD | | X.XX | X.XX | X.XX | X.XX | X.XX |
| Median | | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min. to Max. | | x to x | x to x | x to x | x to x | x to x |
| Oozing and Crusting | | Week 32 | Week 40 | Week 48 | Week 52 | |
| N | | XX | XX | XX | XX | |
| Mean | | X.X | X.X | X.X | X.X | |
| SD | | X.XX | X.XX | X.XX | X.XX | |
| Median | | XX.X | XX.X | XX.X | XX.X | |
| Min. to Max. | | x to x | x to x | x to x | x to x | |
| Change from Baseline | | | | | | |
| N | | XX | XX | XX | XX | |
| Mean | | X.X | X.X | X.X | X.X | |
| SD | | X.XX | X.XX | X.XX | X.XX | |
| Median | | XX.X | XX.X | XX.X | XX.X | |
| Min. to Max. | | x to x | x to x | x to x | x to x | |

Note: No imputation of missing data.

Listing 16.2.7.1

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table 14.3.1.1.2: Means Summary of Local Tolerabilty Reactions by Visit (Safety Population)


| KERYDIN® (N=xx) | | | | | | |
|---|---|---|---|---|---|---|
| Pruritus | Baseline | Week 2 | Week 4 | Week 8 | Week 16 | Week 2 |
| N | XX | XX | XX | XX | XX | XX |
| Mean | X.X | X.X | X.X | X.X | X.X | X.X |
| SD | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min. to Max. | x to x | x to x | x to x | x to x | x to x | x to x |
| Change from Baseline | | | | | | |
| N | | XX | XX | XX | XX | XX |
| Mean | | X.X | X.X | X.X | X.X | X.X |
| SD | | X.XX | X.XX | X.XX | X.XX | X.XX |
| Median | | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min. to Max. | | x to x | x to x | x to x | x to x | x to x |
| Pruritus | | Week 32 | Week 40 | Week 48 | Week 52 | |
| N | | XX | XX | XX | XX | |
| Mean | | X.X | X.X | X.X | X.X | |
| SD | | X.XX | X.XX | X.XX | X.XX | |
| Median | | XX.X | XX.X | XX.X | XX.X | |
| Min. to Max. | | x to x | x to x | x to x | x to x | |
| Change from Baseline | | | | | | |
| N | | XX | XX | XX | XX | |
| Mean | | X.X | X.X | X.X | X.X | |
| SD | | X.XX | X.XX | X.XX | X.XX | |
| Median | | XX.X | XX.X | XX.X | XX.X | |
| Min. to Max. | | x to x | x to x | x to x | x to x | |

Note: No imputation of missing data.

Listing 16.2.7.1

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table 14.3.1.1.2: Means Summary of Local Tolerabilty Reactions by Visit (Safety Population)


| KERYDIN® (N=xx) | | | | | | |
|---|---|---|---|---|---|---|
| Erythema | Baseline | Week 2 | Week 4 | Week 8 | Week 16 | Week 2 |
| N | XX | XX | XX | XX | XX | XX |
| Mean | X.X | X.X | X.X | X.X | X.X | Χ.Σ |
| SD | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min. to Max. | x to x | x to x | x to x | x to x | x to x | x to x |
| Change from Baseline | | | | | | |
| N | | XX | XX | XX | XX | XX |
| Mean | | X.X | X.X | X.X | X.X | х.х |
| SD | | X.XX | X.XX | X.XX | X.XX | X.XX |
| Median | | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min. to Max. | | x to x | x to x | x to x | x to x | x to x |
| Erythema | | Week 32 | Week 40 | Week 48 | Week 52 | |
| N | | XX | XX | XX | XX | |
| Mean | | X.X | X.X | X.X | X.X | |
| SD | | X.XX | X.XX | X.XX | X.XX | |
| Median | | XX.X | XX.X | XX.X | XX.X | |
| Min. to Max. | | x to x | x to x | x to x | x to x | |
| Change from Baseline | | | | | | |
| N | | XX | XX | XX | XX | |
| Mean | | X.X | X.X | X.X | X.X | |
| SD | | X.XX | X.XX | X.XX | X.XX | |
| Median | | XX.X | XX.X | XX.X | XX.X | |
| Min. to Max. | | x to x | x to x | x to x | x to x | |

Note: No imputation of missing data.

Listing 16.2.7.1

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table 14.3.1.1.2: Means Summary of Local Tolerabilty Reactions by Visit (Safety Population)


| KERYDIN® (N=xx) | | | | | | |
|---|---|---|---|---|---|---|
| Scaling | Baseline | Week 2 | Week 4 | Week 8 | Week 16 | Week 24 |
| N | XX | XX | XX | XX | XX | XX |
| Mean | X.X | X.X | X.X | X.X | X.X | X.X |
| SD | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min. to Max. | x to x | x to x | x to x | x to x | x to x | x to x |
| Change from Baseline | | | | | | |
| N | | XX | XX | XX | XX | XX |
| Mean | | X.X | X.X | X.X | X.X | X.X |
| SD | | X.XX | X.XX | X.XX | X.XX | X.XX |
| Median | | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min. to Max. | | x to x | x to x | x to x | x to x | x to x |
| Scaling | | Week 32 | Week 40 | Week 48 | Week 52 | |
| N | | XX | XX | XX | XX | |
| Mean | | X.X | X.X | X.X | X.X | |
| SD | | X.XX | X.XX | X.XX | X.XX | |
| Median | | XX.X | XX.X | XX.X | XX.X | |
| Min. to Max. | | x to x | x to x | x to x | x to x | |
| Change from Baseline | | | | | | |
| N | | XX | XX | XX | XX | |
| Mean | | X.X | X.X | X.X | X.X | |
| SD | | X.XX | X.XX | X.XX | X.XX | |
| Median | | XX.X | XX.X | XX.X | XX.X | |
| Min. to Max. | | x to x | x to x | x to x | x to x | |

Note: No imputation of missing data.

Listing 16.2.7.1

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table 14.3.1.2.1: Summary of Treatment-Emergent Adverse Event Characteristics (Safety Population) 

| | KERYDIN® |
|---|---|
| | (N=xx) |
| Subjects Reporting Any Adverse Event | xx ( xx.x%) |
| Subjects Reporting Any Serious Adverse Event | $XX \left( XX.X^{0}/_{0} \right)$ |
| Subjects Who Died | $XX (XX.X^{0})$ |
| Subjects Who Discontinued Study Drug Due to Adverse Event | xx ( xx.x%) |
| Total Number of Adverse Events Reported | XX |
| By Subject | |
| By Maximum Severity | |
| Mild | xx ( xx.x%) |
| Moderate | xx ( xx.x%) |
| Severe | xx (xx.x%) |
| By Strongest Relationship to Study Drug | $XX \left( XX.X\% \right)$ |
| Definite | xx (xx.x%) |
| Probable | xx ( xx.x%) |
| Possible | xx ( xx.x%) |
| Unlikely | xx (xx.x%) |
| Not Related | xx ( xx.x%) |

Note: Treatment-emergent adverse events are those with an onset on or after the first application of study drug.

Listing 16.2.7.2.3 SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table 14.3.1.2.1: Summary of Treatment-Emergent Adverse Event Characteristics (Safety Population) 

| | KERYDIN® |
|--------------------------------------|-------------|
| | (N=xx) |
| By Subject | |
| Maximum Severity within Relationship | |
| to Study Drug | |
| Definite | |
| Mild | xx ( xx.x%) |
| Moderate | xx ( xx.x%) |
| Severe | xx ( xx.x%) |
| Probable | |
| Mild | xx ( xx.x%) |
| Moderate | xx ( xx.x%) |
| Severe | xx ( xx.x%) |
| Possible | |
| Mild | xx ( xx.x%) |
| Moderate | XX (XX.X%) |
| Severe | xx (xx.x%) |
| Unlikely | |
| Mild | xx (xx.x%) |
| Moderate | xx (xx.x%) |
| Severe | xx (xx.x%) |
| Not Related | |
| Mild | xx (xx.x%) |
| Moderate | XX (XX.X%) |
| Severe | xx (xx.x%) |

Note: Treatment-emergent adverse events are those with an onset on or after the first application of study drug.

Listing 16.2.7.2.3 SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table 14.3.1.2.2: Summary of Treatment-Emergent Adverse Events Leading to Permanent Withdrawal of Study Drug and/or Early Discontinuation From the Study

(Safety Population)

(Page xx of yy)

| System Organ Class <sup>a</sup> Preferred Term | KERYDIN®<br>(N=xx) |
|------------------------------------------------|----------------------------|
| System Organ Class Preferred Term | xx ( xx.x%)<br>xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more adverse events that map to MedDRA. At each level of summarization (System Organ Class or Preferred Term) subjects are counted once.

Note: MedDRA Version 18.0.

Note: Treatment-emergent adverse events are those with an onset on or after the first application of study drug.

Listing 16.2.7.2.3

Table 14.3.1.2.3: Summary of Treatment-Emergent Adverse Events by MedDRA System Organ Class and Preferred Term (Safety Population)

(Page xx of yy)

| System Organ Class <sup>a</sup> Preferred Term | KERYDIN®(N=xx) |
|------------------------------------------------|----------------|
| System Organ Class | xx ( xx.x%) |
| Preferred Term | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more adverse events that map to MedDRA. At each level of summarization (System Organ Class or Preferred Term) subjects are counted once.

Note: MedDRA Version 18.0.

Note: Treatment-emergent adverse events are those with an onset on or after the first application of study drug.

Listing 16.2.7.2.3

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

{NOTE TO PROGRAMMER: Order table by decreasing incidence of Total column. All subsequent tables including summaries by MedDRA SOC and PT should display the SOC and PT in the same order.}

Table 14.3.1.2.4: Summary of Treatment-Emergent Adverse Events by Severity (Safety Population)
(Page xx of yy)

| System Organ Class <sup>a</sup> Preferred Term | <u>Severity</u> | KERYDIN®<br>(N=xx) |
|---|---|---|
| System Organ Class | Mild<br>Moderate<br>Severe | xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%) |
| Preferred Term | Mild<br>Moderate<br>Severe | xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more adverse events that map to MedDRA. At each level of summarization (System Organ Class or Preferred Term) subjects are counted once under the greatest reported severity.

Note: MedDRA Version 18.0.

Note: Treatment-emergent adverse events are those with an onset on or after the first application of study drug.

Listing 16.2.7.2.3

Table 14.3.1.2.4: Summary of Treatment-Emergent Adverse Events by Relationship (Safety Population)
(Page xx of yy)

| System Organ Class <sup>a</sup> Preferred Term | <u>Relationship</u> | KERYDIN®<br>(N=xx) |
|---|---|---|
| System Organ Class | Definite<br>Probable<br>Possible<br>Unlikely<br>Not Related | xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%) |
| Preferred Term | Definite<br>Probable<br>Possible<br>Unlikely<br>Not Related | xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more adverse events that map to MedDRA. At each level of summarization (System Organ Class or Preferred Term) subjects are counted once under the greatest reported relationship.

Note: MedDRA Version 18.0.

Note: Treatment-emergent adverse events are those with an onset on or after the first application of study drug.

Listing 16.2.7.2.3

Table 14.3.2.2.1: Summary of Treatment-Emergent Serious Adverse Event Characteristics (Safety Population)


| Subjects Reporting Any Serious Adverse Event<br>Subjects Who Died<br>Subjects Who Discontinued Study Drug Due to Adverse Event | KERYDIN® |
|---|---|
| Total Number of Adverse Events Reported | XX |
| By Subject By Maximum Severity Mild Moderate Severe | xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%) |
| By Strongest Relationship to Study Drug Definite Probable Possible Unlikely Not Related | xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%) |

Note: Treatment-emergent serious adverse events are those with an onset on or after the first application of study drug.

Listing 16.2.7.2.4

Table 14.3.2.2.1: Summary of Treatment-Emergent Serious Adverse Event Characteristics (Safety Population) 

| | KERYDIN® |
|--------------------------------------|-------------|
| | (N=xx) |
| By Subject | |
| Maximum Severity within Relationship | |
| to Study Drug | |
| Definite | |
| Mild | xx ( xx.x%) |
| Moderate | xx ( xx.x%) |
| Severe | xx ( xx.x%) |
| Probable | |
| Mild | xx ( xx.x%) |
| Moderate | xx ( xx.x%) |
| Severe | xx ( xx.x%) |
| Possible | |
| Mild | xx ( xx.x%) |
| Moderate | xx ( xx.x%) |
| Severe | xx ( xx.x%) |
| Unlikely | |
| Mild | xx ( xx.x%) |
| Moderate | xx ( xx.x%) |
| Severe | xx ( xx.x%) |
| Not Related | |
| Mild | xx ( xx.x%) |
| Moderate | xx ( xx.x%) |
| Severe | xx ( xx.x%) |

Note: Treatment-emergent serious adverse events are those with an onset on or after the first application of study drug.

Listing 16.2.7.2.4 SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table 14.3.2.2.2: Summary of Treatment-Emergent Serious Adverse Events by MedDRA System Organ Class and Preferred Term (Safety Population)

(Page xx of yy)

| System Organ Class <sup>a</sup> Preferred Term | KERYDIN®<br>(N=xx) |
|------------------------------------------------|----------------------------|
| System Organ Class Preferred Term | xx ( xx.x%)<br>xx ( xx.x%) |

Note: MedDRA Version 18.0.

Note: Treatment-emergent serious adverse events are those with an onset on or after the first application of study drug.

Listing 16.2.7.2.4

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more serious adverse events that map to MedDRA. At each level of summarization (System Organ Class or Preferred Term) subjects are counted once.

Table 14.3.2.2.3: Summary of Treatment-Emergent Serious Adverse Events by Severity (Safety Population)
(Page xx of yy)

| System Organ Class <sup>a</sup> Preferred Term | <u>Severity</u> | KERYDIN®<br>(N=xx) |
|---|---|---|
| System Organ Class | Mild<br>Moderate<br>Severe | xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%) |
| Preferred Term | Mild<br>Moderate<br>Severe | xx ( xx.x%)<br>xx ( xx.x%)<br>xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more serious adverse events that map to MedDRA. At each level of summarization (System Organ Class or Preferred Term) subjects are counted once under the greatest reported severity.

Note: MedDRA Version 18.0.

Note: Treatment-emergent serious adverse events are those with an onset on or after the first application of study drug.

Listing 16.2.7.2.4

Table 14.3.2.2.4: Summary of Treatment-Emergent Serious Adverse Events by Relationship (Safety Population)

(Page xx of yy)

| System Organ Class <sup>a</sup> | | <b>KERYDIN®</b> |
|---------------------------------|---------------------|-----------------|
| Preferred Term | <u>Relationship</u> | (N=xx) |
| System Organ Class | Definite | xx ( xx.x%) |
| | Probable | xx ( xx.x%) |
| | Possible | xx ( xx.x%) |
| | Unlikely | xx ( xx.x%) |
| | Not Related | xx ( xx.x%) |
| Preferred Term | Definite | xx ( xx.x%) |
| | Probable | xx ( xx.x%) |
| | Possible | xx ( xx.x%) |
| | Unlikely | xx ( xx.x%) |
| | Not Related | xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects reporting one or more serious adverse events that map to MedDRA. At each level of summarization (System Organ Class or Preferred Term) subjects are counted once under the greatest reported relationship.

Note: MedDRA Version 18.0.

Note: Treatment-emergent serious adverse events are those with an onset on or after the first application of study drug.

Listing 16.2.7.2.4

Table 14.3.4.1.1: Summary of Hematology Results (Safety Population)
(Page 1 of x)

| | | KERYDIN®<br>(N=xxx) | | | | | |
|---|---|---|---|---|---|---|---|
| Test name (units) | | | | CI C | | | CI C |
| | | Baseline | Week 24 | Change from Baseline | Baseline | Week 52 | Change from Baseline |
| N | | XXX | Xxx | XXX | XXX | XXX | XXX |
| Mean | | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | | XX.XX | XX.XX | XX.XX | XX,XX | XX.XX | XX.XX |
| Median | | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min. to Max. | | xx to xx | xx to xx | xx to xx | xx to xx | xx to xx | xx to xx |
| | | | Week 24 | | | Week 52 | |
| | <b>Baseline</b> | BNL | WNL | ANL | BNL | WNL | ANL |
| | BNL | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | WNL | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | ANL | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

Note: BNL=Below Normal Limit, WNL=Within Normal Limits, ANL=Above Normal Limit.

Note: No imputation of missing values.

Listing 16.2.8.2.1

Table 14.3.4.1.2: Summary of Chemistry Results (Safety Population)
(Page 1 of x)

| | | KERYDIN® (N=xxx) | | | | | |
|---|---|---|---|---|---|---|---|
| Test name (units) | | | | | | | |
| | | | | Change from | | | Change from |
| | | Baseline | Week 24 | Baseline | Baseline | Week 52 | Baseline |
| N | | XXX | XXX | XXX | XXX | XXX | XXX |
| Mean | | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min. to Max. | | xx to xx | xx to xx | xx to xx | xx to xx | xx to xx | xx to xx |
| | | | Week 24 | | | Week 52 | |
| | <b>Baseline</b> | BNL | WNL | ANL | BNL | WNL | ANL |
| | BNL | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) | xx (xx.x%) | xx ( xx.x%) |
| | WNL | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | ANL | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

Note: BNL=Below Normal Limit, WNL=Within Normal Limits, ANL=Above Normal Limit.

Listing 16.2.8.2.1

Table 14.3.5.1: Summary of Vital Signs by Visit (Safety Population)


| KERYDIN® (N=xx) | | | | | | |
|---|---|---|---|---|---|---|
| Systolic Blood Pressure (mmHg) | Baseline | Week 2 | Week 4 | Week 8 | Week 16 | Week 24 |
| N | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX,XX | XX.XX | XX.XX | XX.XX | XX,XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | | | | |
| N | | XX | XX | XX | XX | XX |
| Mean | | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min. to Max. | | xx to xx | xx to xx | xx to xx | xx to xx | xx to xx |
| Systolic Blood Pressure (mmHg) | | Week 32 | Week 40 | Week 48 | Week 52 | |
| N | | XX | XX | XX | XX | |
| Mean | | XX.X | XX.X | XX.X | XX.X | |
| SD | | XX.XX | XX.XX | XX.XX | XX.XX | |
| Median | | XX.X | XX.X | XX.X | XX.X | |
| Min. to Max. | | xx to xx | xx to xx | xx to xx | xx to xx | |
| Change from Baseline | | | | | | |
| N | | XX | XX | XX | XX | |
| Mean | | XX.X | XX.X | XX.X | XX.X | |
| SD | | XX.XX | XX.XX | XX.XX | XX.XX | |
| Median | | XX.X | XX.X | XX.X | XX.X | |
| Min. to Max. | | xx to xx | xx to xx | xx to xx | xx to xx | |

Note: No imputation of missing data.

Listing16.2.8.3

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table 14.3.5.1: Summary of Vital Signs by Visit (Safety Population)


| KERYDIN® (N=xx) | | | | | | |
|---|---|---|---|---|---|---|
| Diastolic Blood Pressure (mmHg) | Baseline | Week 2 | Week 4 | Week 8 | Week 16 | Week 24 |
| N | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | | | | |
| N | | XX | XX | XX | XX | XX |
| Mean | | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min. to Max. | | xx to xx | xx to xx | xx to xx | xx to xx | xx to xx |
| Diastolic Blood Pressure (mmHg) | | Week 32 | Week 40 | Week 48 | Week 52 | |
| N | | XX | XX | XX | XX | |
| Mean | | XX.X | XX.X | XX.X | XX.X | |
| SD | | XX.XX | XX.XX | XX.XX | XX.XX | |
| Median | | XX.X | XX.X | XX.X | XX.X | |
| Min. to Max. | | xx to xx | xx to xx | xx to xx | xx to xx | |
| Change from Baseline | | | | | | |
| N | | XX | XX | XX | XX | |
| Mean | | XX.X | XX.X | XX.X | XX.X | |
| SD | | XX.XX | XX.XX | XX.XX | XX.XX | |
| Median | | XX.X | XX.X | XX.X | XX.X | |
| Min. to Max. | | xx to xx | xx to xx | xx to xx | xx to xx | |

Note: No imputation of missing data.

Listing16.2.8.3

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table 14.3.5.1: Summary of Vital Signs by Visit (Safety Population)


| KERYDIN® (N=xx) | | | | | | |
|---|---|---|---|---|---|---|
| Pulse Rate (beats/min) | Baseline | Week 2 | Week 4 | Week 8 | Week 16 | Week 24 |
| N | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | | | | |
| N | | XX | XX | XX | XX | XX |
| Mean | | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min. to Max. | | xx to xx | xx to xx | xx to xx | xx to xx | xx to xx |
| Pulse Rate (beats/min) | | Week 32 | Week 40 | Week 48 | Week 52 | |
| N | | XX | XX | XX | XX | |
| Mean | | XX.X | XX.X | XX.X | XX.X | |
| SD | | XX.XX | XX.XX | XX.XX | XX.XX | |
| Median | | XX.X | XX.X | XX.X | XX.X | |
| Min. to Max. | | xx to xx | xx to xx | xx to xx | xx to xx | |
| Change from Baseline | | | | | | |
| N | | XX | XX | XX | XX | |
| Mean | | XX.X | XX.X | XX.X | XX.X | |
| SD | | XX.XX | XX.XX | XX.XX | XX.XX | |
| Median | | XX.X | XX.X | XX.X | XX.X | |
| Min. to Max. | | xx to xx | xx to xx | xx to xx | xx to xx | |

Note: No imputation of missing data.

Listing16.2.8.3

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table 14.3.5.1: Summary of Vital Signs by Visit (Safety Population)


| KERYDIN® (N=xx) | | | | | | |
|---|---|---|---|---|---|---|
| Respiratory Rate (breaths/min) | Baseline | Week 2 | Week 4 | Week 8 | Week 16 | Week 24 |
| N | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx | xx to xx | xx to xx | xx to xx |
| Change from Baseline | | | | | | |
| N | | XX | XX | XX | XX | XX |
| Mean | | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min. to Max. | | xx to xx | xx to xx | xx to xx | xx to xx | xx to xx |
| Respiratory Rate (breaths/min) | | Week 32 | Week 40 | Week 48 | Week 52 | |
| N | | XX | XX | XX | XX | |
| Mean | | XX.X | XX.X | XX.X | XX.X | |
| SD | | XX.XX | XX.XX | XX.XX | XX.XX | |
| Median | | XX.X | XX.X | XX.X | XX.X | |
| Min. to Max. | | xx to xx | xx to xx | xx to xx | xx to xx | |
| Change from Baseline | | | | | | |
| N | | XX | XX | XX | XX | |
| Mean | | XX.X | XX.X | XX.X | XX.X | |
| SD | | XX.XX | XX.XX | XX.XX | XX.XX | |
| Median | | XX.X | XX.X | XX.X | XX.X | |
| Min. to Max. | | xx to xx | xx to xx | xx to xx | xx to xx | |

Note: No imputation of missing data.

Listing16.2.8.3

SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Table 14.4.1: Extent of Exposure (Safety Population)

| | KERYDIN® |
|----------------------------------------|----------|
| | (N=xx) |
| Total Number of Dosing Days | |
| N | XX |
| Mean | XX.X |
| SD | XX.XX |
| Median | XX.X |
| Min. to Max. | xx to xx |
| Total Number of Applications | |
| N | XX |
| Mean | XX.X |
| SD | XX.XX |
| Median | XX.X |
| Min. to Max. | xx to xx |
| Total Amount of Study Drug Applied (g) | |
| N | XX |
| Mean | XX.X |
| SD | XX.XX |
| Median | XX.X |
| Min. to Max. | xx to xx |

Listings 16.2.5.2, 16.2.5.3

# Table 14.4.2: Summary of Concomitant Medications (Safety Population) (Page xx of yy)

| ATC Level 2 Term <sup>a</sup> Preferred Name | KERYDIN®(N=xx) |
|----------------------------------------------|----------------------------|
| ATC Level 2 Term Preferred Name | xx ( xx.x%)<br>xx ( xx.x%) |

<sup>&</sup>lt;sup>a</sup> Counts reflect numbers of subjects with concomitant medications that map to WHO-DDE. At each level of summarization (ATC Level 2 Term or Preferred Name) subjects are counted once.

Note: WHO-DDE Format B2, Version March 1, 2015.

Listing 16.2.4.3.2

Table 14.4.4.1: Summary of Tavaborole Plasma Concentrations (PK Population)

| KERYDIN® (N=xx) | | | Day 15 | | |
|---|---|---|---|---|---|
| | Pre-Dose | | • | | |
| Plasma Concentration | | | | | |
| Below the Lower Limit of Quantification | xxx ( xx.x%) | | | | |
| Detectable Concentrations | | | | | |
| N | XXX | | | | |
| Mean | XX.X | | | | |
| SD | XX.XX | | | | |
| Median | XX.X | | | | |
| Min. to Max. | xx to xx | | | | |
| | | | Day 29 | | |
| | Pre-Dose | 4 Hour Post-Dose | 6 Hours Post-Dose | 8 Hours Post-Dose | 24 Hours Post-Dose |
| Plasma Concentration | | | | | |
| Below the Lower Limit of Quantification | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Detectable Concentrations | | | | | |
| N | XXX | XXX | XXX | XXX | XXX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min. to Max. | xx to xx | xx to xx | xx to xx | xx to xx | xx to xx |

Note: Lower Limit of Quantification = x ng/mL

Note: No imputation of missing data.

Listing 16.2.6.3 SOURCE: USERNAME\SPONSOR\PROJECT\JOBNAME (DATE,TIME)

Figure 14.4.4.1.1: Linear Plot of Mean Plasma Concentrations of Tavaborole by Time (PK Population)
(Page xx of yy)



Note: Figure represents mean concentrations +/- standard errors.

Note: No imputation of missing data.

Figure 14.4.4.1.2: Semi-logarithmic Plot of Mean Plasma Concentrations of Tavaborole by Time (PK Population)
(Page xx of yy)



Note: Figure represents mean concentrations +/- standard errors.

Note: No imputation of missing data.

Figure 14.4.4.1.3: By-Subject Linear Plots of Plasma Concentrations of Tavaborole by Time (PK Population)
(Page xx of yy)



Note: No imputation of missing data.

Figure 14.4.4.1.4: By-Subject Semi-logarithmic Plots of Plasma Concentrations of Tavaborole by Time (PK Population)
(Page xx of yy)



Note: No imputation of missing data.

Table 14.4.5.1: Summary of Pharmacokinetic Parameters of Tavaborole at Day 29 (PK Population)


| | KERYDIN® |
|---------------------------|---------------------------------------|
| Day 29 | N=xx |
| C | · |
| Day 29 C <sub>max</sub> N | XX |
| Mean | XX,X |
| SD | |
| | XX.XX |
| Median | XX.X |
| Min. to Max. | xx to xx |
| $T_{\text{max}}$ | |
| N | XX |
| Mean | XX.X |
| SD | XX.XX |
| Median | XX.X |
| Min. to Max. | xx to xx |
| $AUC_{0-24}$ | |
| N | XX |
| Mean | |
| | XX.X |
| SD | XX.XX |
| Median | XX.X |
| Min. to Max. | xx to xx |

Note: Lower Limit of Quantification = x ng/mL

Note: No imputation of missing data.

Listing 16.2.6.4

Table 14.4.5.1: Summary of Pharmacokinetic Parameters at Day 29 (PK Population) 

| | KERYDIN® |
|------------------------------------------|----------|
| Day 29 | (N=xx) |
| $\mathrm{AUC}_{0\text{-}\infty}$ | |
| N | XX |
| Mean | XX.X |
| SD | XX.XX |
| Median | XX.X |
| Min. to Max. | xx to xx |
| Constant of Elimination ( $\lambda_Z$ ) | |
| N | XX |
| Mean | XX.X |
| SD | XX.XX |
| Median | XX.X |
| Min. to Max. | xx to xx |
| Elimination half-life (t <sub>1/2)</sub> | |
| N | XX |
| Mean | XX.X |
| SD | XX.XX |
| Median | XX.X |
| Min. to Max. | xx to xx |

Note: Lower Limit of Quantification = x ng/mL

Note: No imputation of missing data.

Listing 16.2.6.4

# 7. INDEX OF PLANNED LISTINGS